CLINICAL TRIAL: NCT04657640
Title: Scaling-up High-impact Micronutrient Supplementation Interventions to Improve Adolescents' Nutrition and Health in Burkina Faso
Brief Title: School-Based Assessment of Micronutrient Interventions in Adolescents in Burkina Faso
Acronym: SAMIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Centre de Recherche en Sante de Nouna, Burkina Faso (Other Government)
Responsible Party: Principal Investigator, Wafaie Fawzi, Professor of Nutrition, Epidemiology, and Global Health, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB20-1108
Record Dates: First submitted 2020-11-24; First posted 2020-12-08 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Anemia
Keywords: Multiple Micronutrient Supplementation; Iron and Folic Acid; Nutrition; Adolescent Health
MeSH Terms: conditions — Anemia | interventions — Iron; Folic Acid

STUDY DESIGN:
Intervention Model Description: Schools will be randomly assigned to weekly iron and folic acid (IFA) supplementation; daily multiple micronutrient supplements (MMS); or control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- weekly iron and folic acid supplementation (IFA) (Experimental)
  Interventions: Dietary Supplement: Iron and folic acid (IFA)
- daily multiple micronutrient supplement (MMS) (Experimental)
  Interventions: Dietary Supplement: Multiple Micronutrient Supplements (MMS) and loading dose of Iron and Folic Acid (IFA)
- control (No Intervention)

INTERVENTIONS:
Dietary Supplement: Iron and folic acid (IFA) — Weekly regimen of one tablet containing Iron (60mg) and Folic Acid (2800 μg) for 3 months intermittently
  Arms: weekly iron and folic acid supplementation (IFA)
Dietary Supplement: Multiple Micronutrient Supplements (MMS) and loading dose of Iron and Folic Acid (IFA) — Daily regimen of MMS for 3 months intermittently. MMS is the United Nations International Multiple Micronutrient Antenatal Preparation (UNIMMAP) tablet containing fifteen micronutrients including iron (30mg), folic acid (400 mcg), Vit A, Retinol (800 RE), vit D (200 IU), vit E (10 mg), vit C (70 mg), vit B1 (1.4 mg), vit B2 (1.4 mg), vit B6 (1.9 mg), vit B12 (2.6 mcg), niacin (18 mg), zinc (15 mg), copper (2 mg), iodine (150 mcg), selenium (65 mcg).
  For the first 5 weeks of the study, participants will also receive weekly regimen of one tablet containing Iron (60mg) and Folic Acid (2800 μg) as a loading dose, in addition to daily MMS.
  Arms: daily multiple micronutrient supplement (MMS)

SUMMARY:
This purpose of this study is to assess effects of iron and folic acid supplementation and multiple micronutrient supplementation on anemia status, school performance/attendance and development outcomes among adolescents in Burkina Faso.

DETAILED DESCRIPTION:
This study aims to implement and evaluate micronutrient supplementation interventions to improve adolescent nutrition, health and education in Burkina Faso. Findings from this study will clarify the optimal supplementation strategy (iron and folic acid alone or adding other essential nutrients) and provide a basis for scale up of national micronutrient supplementation programs to benefit the adolescent population as a whole in Burkina Faso.

This will be a cluster randomized study with 3 arms. 42 schools per country will be enrolled (14 schools per arm) to receive either 1) daily Multiple Micronutrient Supplements (MMS) and weekly Iron and Folic Acid (IFA) for the first 5 weeks and daily MMS for the remainder of the study; or 2) weekly IFA; or 3) to serve as controls. As recommended by the World Health Organization in settings where continuous supplementation is not possible, supplementation will be intermittent. Supplementation will be provided for 3 months, stopped for 3 months over the school summer holidays and resumed for 3 months once students return to school after the holiday. Students in intervention schools will receive supplementation and students in control schools will receive the usual care (which does not include supplementation but does include existing curriculum on nutrition and water, sanitation and hygiene [WASH]). The program will be evaluated comparing effects of weekly IFA and daily MMS on anemia status and school attendance/retention.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 10-17 years
* Enrolled in secondary school form 1 at study initiation
* Member of one of the selected classes in a participating school
* Consent provided by the parent
* Assent provided by the adolescent
* Fluency in French

Exclusion Criteria:

* No informed consent from parent or assent from adolescent
* Self-reported Pregnancy

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3123 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Anemia Status | Up to one year
  Anemia will be defined as hemoglobin level <10 g/dL

SECONDARY OUTCOMES:
School attendance | Up to one year
  School attendance will be measured as number of days of missed school per student
School retention | Up to one year
  School retention will be measured as number of students who drop out of school

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Wafaie, MBBS, MPH, MS, DrPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Nouna Health Research Center, Nouna, Burkina Faso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cliffer IR, Millogo O, Barry Y, Kouanda I, Compaore G, Wang D, Sie A, Fawzi W. School-based supplementation with iron-folic acid or multiple micronutrient tablets to address anemia among adolescents in Burkina Faso: a cluster-randomized trial. Am J Clin Nutr. 2023 Nov;118(5):977-988. doi: 10.1016/j.ajcnut.2023.09.004. Epub 2023 Sep 15. PMID 37716443
- [Derived] Cliffer IR, Yussuf MH, Millogo O, Mwanyika-Sando M, Barry Y, Yusufu IS, Hemler EC, Sie A, Tinkasimile A, Compaore G, Ali AS, Kouanda I, Wang D, Mosha D, Fawzi W. Scaling-up high-impact micronutrient supplementation interventions to improve adolescents' nutrition and health in Burkina Faso and Tanzania: protocol for a cluster-randomised controlled trial. BMJ Open. 2023 Feb 15;13(2):e063686. doi: 10.1136/bmjopen-2022-063686. PMID 36792333